CLINICAL TRIAL: NCT00979095
Title: Genetic Differences Between Patients With Multiple Hernia and a Healthy Control Group
Brief Title: Genetic Examination of Patients With Primary Multiple Hernia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Jakob Burcharth, MD., Herlev Hospital
Other Study IDs: H-D-2008-126
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Multiple Hernia
Keywords: multiple hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple hernia: Patients with more than 3 primary hernias
- Control group: Patients without hernias

SUMMARY:
The investigators are performing a genetic study of patients with multiple hernias (at least 3 primary hernias) versus a healthy control group. This genetic information is compared with circulating and subcutaneously biomarkers such as matrix-metalloproteinases (MMP's).

The hypothesis is that patients with multiple hernias have different expression of specific genes compared to the healthy control group.

DETAILED DESCRIPTION:
Other examinations performed on the patients enrolled in this study:

* Ultrasound (US) examination of the abdominal aorta to discover possible abdominal aortic aneurysms.
* Beightons score to evaluate the degree of joint hypermobility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with minimum 3 primary hernias

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish citizens. Data have been retracted from The Danish Hernia Database.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Genetic expression of relevant genes between the groups | 12 months

SECONDARY OUTCOMES:
Amount of serological biomarkers (MMP's) correlated to gene expression | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Prof. MD, Study Director — Herlev Hospital; Jakob Burcharth, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Jacob Rosenberg, Herlev Hospital, Herev, Denmark